CLINICAL TRIAL: NCT00713271
Title: A Phase I, Randomised, Double-blind, Placebo-controlled, Parallel-group, Single-centre Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of AZD3199 (a B2-agonist) Given Once Daily as Inhaled Formulation Via Turbuhaler to Healthy Men
Brief Title: Multiple Ascending Doses (MAD) of AZD3199 Given Once Daily as Inhaled Formulation Via Turbuhaler to Healthy Men
Acronym: AZD3199MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0570C00002
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy male; tolerability; safety; inhalation
MeSH Terms: conditions — Respiratory Aspiration | interventions — AZD-3199

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Low dose
  Interventions: Drug: AZD3199
- 2 (Experimental): intermediate dose
  Interventions: Drug: AZD3199
- 3 (Experimental): high dose
  Interventions: Drug: AZD3199
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3199 — Low dose
  Dry powder for inhalation, o.d., 1+12 days
  Arms: 1
Drug: Placebo
  Arms: 4
Drug: AZD3199 — intermediate dose
  Dry powder for inhalation, o.d., 1+12 days
  Arms: 2
Drug: AZD3199 — high dose
  Dry powder for inhalation, o.d., 1+12 days
  Arms: 3

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of multiple once daily ascending doses of AZD3199 in healthy men

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-30, weight 60-100 kg
* Non/ex-smokers, Non/ex-nicotine users

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically relevant abnormal findings at screening examinations
* Use of any prescribed or non-prescribed medication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of Adverse Events | Before, during and after dosing
Clinical significant abnormalities in ECG, pulse, blood pressure, lung function, temp, lab | Before, during and after dosing

SECONDARY OUTCOMES:
Pharmacokinetics | Before, during and after dosing
Potassium and lactate concentrations | Before, during and after dosing
Tremor, palpitations, heart rate, QTc, pulse and blood pressure and FEV1 | Before, during and after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Samuelsson Palmgren, Principal Investigator — AZ CPU Lund, Sweden
Locations (1):
- Research Site, Lund, Sweden

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1662&filename=CSR-D0570C00002.pdf
- See also: CSR-D0570C00002.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1662&filename=CSR-D0570C00002.pdf